CLINICAL TRIAL: NCT05613881
Title: The Effect of Education and Telephone Follow-up on Quality of Life and Symptom Management in Patients Receiving Androgen Deprivation Therapy
Brief Title: Symptom Management, Education and Telephone Follow-up, Quality of Life,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Prof. Dr. Ayfer ÖZBAŞ (Unknown)
Responsible Party: Principal Investigator, Tuğba Sınmaz, RESEARCH ASSISTANT MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-74555795-050.01.04-185078
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Deprivation Therapy; Telephone Follow-up; Nursing Education
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Experimental and control groups will be formed by randomization from individuals who meet the inclusion criteria. At the beginning of the research, a pre-test will be applied to both groups at the first interview. The individuals in the experimental group will be given an education and training booklet prepared in line with the literature by the researcher at the first interview. Only the training booklet will be given to the control group. Individuals in the experimental group will be called every 15 days for 3 months, in line with the Telephone Monitoring Instruction Form, to be interviewed and monitored. At the end of the 3rd month, the final tests will be applied. Individuals in the control group will be given post-tests at the end of the 3rd month..
Who Masked: Participant
Masking Description: The participant does not know which group he is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): the group to be trained and then monitored by phone
  Interventions: Other: Education and Telephone Follow-up
- CONTROL GROUP (No Intervention): The individuals in this group will be given only education booklet by the researcher after the pre-tests are applied in the first face-to-face interview. 3 months after the first interview, the final tests will be applied.

INTERVENTIONS:
Other: Education and Telephone Follow-up — The individuals in this group will be given an education and training booklet by the researcher after the pre-tests are applied in the first face-to-face interview. After the first meeting, the individual will be called every 15 days, 5 times in total for 3 months, and the training will be repeated in line with the individual's needs. After 3 months, the final tests will be applied.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
This study was planned as an experimental design study with pretest-posttest control group in order to determine the effects of education and telephone follow-up given to patients receiving androgen deprivation therapy (ADT) for prostate cancer on quality of life and symptom management.The main question[s] it aims to answer are:

* Is the quality of life higher in patients receiving androgen deprivation therapy who are trained and followed up over the phone compared to patients who are only given an education booklet?
* Is symptom management higher in patients receiving androgen deprivation therapy who received training and followed-up over the phone compared to patients who were only given an education booklet?

DETAILED DESCRIPTION:
The number of samples to be taken in each group was determined as 24 (total 48) with the help of the G-power (version 3.1) package program. Considering the possible losses in the research and in order to increase the power of the study, it was planned to carry out the research with a total of 60 people, 30 people in the experimental and control groups.

While evaluating the findings obtained in the study, SPSS (Statistical Package for the Social Sciences) version 25.0 (IBM Corp., Armonk, NY, USA) program will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Literate and open to communication,
* Knowing the diagnosis,
* Those aged 45 and over,
* Receiving short-term or long-term ADT treatment,
* The patient or his/her relatives have telephone access,

Exclusion Criteria:

* Having a mental or psychiatric illness that prevents communication,
* Those with vision-hearing problems

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-C30 (Version 3.0) Quality of Life Scale | Through study completion, an average of 3 months
  It is a questionnaire to measure quality of life which consists of three parts, namely "General Health Status Scale", "Functional Scale", "Symptom Scale" and a total of 30 questions. The last two questions (29,30); provides an assessment of the global quality of life. Each item in the scale is evaluated between 0 and 100 points. For each of the 28 questions in the functional scale and symptom scale, there are four options as none (1 point), a little (2 points), quite (3 points), a lot (4 points). On the general health scale, there are options ranging from very bad to excellent in the range of 1-7 points. Higher values represent a better situation
EORTC QLQ-PR25 Prostate Module | Through study completion, an average of 3 months
  It is a questionnaire to measure quality of life and consisting of 25 items. Prostate Cancer-specific side effects related to surgery, radiotherapy or hormonal therapy that are not in QLQ-C30; voiding problems, bowel functions, sexual status. It consists of two functional (sexual activity and sexual function) and four symptom scales (urinary, intestinal, hormone therapy-related symptoms and incontinence). The score of each item in the scale is evaluated by converting it into a linear range of 0 to 100 points. For each of the 25 questions in the module, there are four options: none (1 point), a little (2 points), quite (3 points), a lot (4 points). A high score from the functional scale indicates a high functional level, and a high score from the symptom scale indicates that the symptoms are experienced intensely.

SECONDARY OUTCOMES:
The blood pressure measurements | 3 months
  Blood pressure monitoring will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Blood pressure measurement is performed by the researcher using the same manual sphygmomanometer instrument during pretest and posttest data collection. Blood pressure is expressed in "mmHg".
The heart rate measurement | 3 months
  Heart rate monitoring will be used to evaluate metabolic and cardiovascular risk factors, whichis side effect of ADT. The heart rate is measured by the researcher by counting over the radial artery for one minute during pretest and posttest data collection. Heart rate refers to the number of beats per minute.
Weight | 3 months
  Weight monitoring will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Weight measurement is performed by the researcher using the wall weight meter during pretest and posttest data collection. Weight is expressed in "kilograms".
Height | 3 months
  Height monitoring will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Height measurement is performed by the researcher using wall height meter during pretest and posttest data collection. Height is expressed in "meters".
BMI | 3 months
  BMI monitoring will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Weight and height will be combined to report BMI in kg/m^2.
Waist/Hip circumference measurement | 3 months
  Waist/Hip circumference measurement will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Waist circumference/hip circumference is measured with a plastic flexible tape measure while the patient is standing in an upright position. Waist/Hip circumference measurement is expressed in "centemeter".
Prostate Spesific Antigen (PSA) | 3 months
  Prostate Specific Antigen (PSA) parameter will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Prostate Specific Antigen (PSA) will be obtained from the hospital automation system during pretest and posttest data collection. PSA is expressed in "(nanogram/milliliter) ng/ml".
Glucose level | 3 months
  Glucose levels parameter will be used to evaluate metabolic and cardiovascular risk factors, which is side effect of ADT. Glucose level will be obtained from the hospital automation system during pretest and posttest data collection. Glucose level is expressed in "(milligram/deciliter) mg/dl".

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No